CLINICAL TRIAL: NCT07058181
Title: A Meaning-centered Intervention for Individuals Who Tend to Feel Down or Anxious
Brief Title: Meaning-centered Intervention for Internalizing Symptoms
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: University of Groningen (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PSY-2324-S-0451; Gravitation 024.004.016 (Other Grant/Funding Number: NWO)
Record Dates: First submitted 2025-05-16; First posted 2025-07-10 (Actual); Last update posted 2025-07-10 (Actual); Status verified 2025-05

CONDITIONS: Depressive and/or Anxiety Symptoms
Keywords: meaning-centered intervention; internalizing symptoms; young adults

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Meaning-centered intervention (Experimental): Participants receive a meaning-centered intervention consisting of six 1-hour online sessions led by a trainer.
  Interventions: Behavioral: Meaning-centered intervention for individuals who tend to feel down or anxious
- Waitlist control (No Intervention): No task or intervention is assigned to participants in this arm.

INTERVENTIONS:
Behavioral: Meaning-centered intervention for individuals who tend to feel down or anxious — Meaning-centered intervention for internalizing symptoms adapted from the intervention "Meaning-centered intervention for youth worrying about their weight and shape".
  * Six 1-hour individual online sessions, approximately every 4 days
  * Sessions led by a certified trainer based on intervention manual
  * Four sources of meaning will be explored: personal life story, dealing with life's limitations, creating one's own life, and meaningful experiences
  * Participants follow intervention using intervention workbook
  * Homework assignments designed to deepen participants' experience and reflection on meaning in their daily lives
  Arms: Meaning-centered intervention

SUMMARY:
Young adults with internalizing symptoms will be randomly assigned to a six-session meaning-centered intervention condition or a waitlist condition. Both conditions receive the same questionnaires at baseline, post assessment (intervention condition: immediately after the final session; waitlist: four weeks after baseline), and follow-up.

The researchers hypothesize that a meaning-centered intervention for individuals with internalizing symptoms will increase participants' meaning in life and reduce their internalizing symptoms at post assessment and 4-week follow-up when compared to a waitlist condition.

DETAILED DESCRIPTION:
First-year psychology students at the University of Groningen will be screened for depressive and anxiety symptoms. Those with heightened symptoms will be invited via e-mail to participate in the study. After filling out the baseline assessment online, participants will be randomly assigned to either a meaning-centered intervention condition, which will receive a meaning-centered intervention taking place approximately every four days, or a waitlist condition, which will be assigned no task. Participants in the intervention condition will follow six 1-hour online intervention sessions led by a trainer and conduct intervention-related homework assignments. The sessions can be followed in English, Dutch, or German. The intervention aims to increase participants' meaning in life and reduce their internalizing symptoms (i.e. depressive and/or anxiety symptoms). Immediately after the final session (i.e. approximately one month after the baseline assessment), participants in the intervention condition will be asked to fill in the post assessment, which includes the same questionnaires as the baseline assessment. Participants in the waitlist control will be asked to complete the post assessment one month after their baseline assessment. One month after the post assessment, participants in both conditions are asked to fill in same set of questionnaires. Waitlist participants are offered to receive the intervention sessions after the study has finished. Participants are compensated with SONA credits.

ELIGIBILITY:
Inclusion Criteria:

* heightened internalizing symptoms (depressive and/or anxiety symptoms) as indicated by PHQ-4 total score of 2 or higher

Exclusion Criteria:

* receiving psychotherapeutic treatment for a depressive or anxiety disorder
* suicidality

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 142 (Estimated)
Dates: Start 2024-11-28 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Meaning in Life Questionnaire; Depression, Anxiety and Stress Scales-21 | at baseline; post (one month after baseline); one-month follow-up (one month after post)
  questionnaire (MLQ: sum score (5-35), 7-point Likert scale (1-7), higher scores indicating higher presence of life meaning; DASS-21: sum score (0-33), 4-point Likert scale (0-3), higher scores indicating higher internalizing symptoms)

SECONDARY OUTCOMES:
Dyscontrolled drinking; Three-dimensional meaning | at baseline; post (one month after baseline); one-month follow-up (one month after post)
  questionnaire (Dyscontrolled drinking: sum score (3-27), 9-point Likert scale (1-9), higher scores indicating higher dyscontrolled drinking; Three-dimensional meaning: sum score (11-77), 7-Point Likert scale (1-7), higher scores indicating higher life meaning)

CONTACTS AND LOCATIONS:
Locations (1):
- Heymans Institute, Groningen, Netherlands

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2025-06-19): https://cdn.clinicaltrials.gov/large-docs/81/NCT07058181/Prot_SAP_ICF_000.pdf